CLINICAL TRIAL: NCT00459719
Title: A Multicenter, Randomized, Open Label, Parallel Study to Evaluate and Compare the Efficacy and Safety of FK506MR vs Prograf® in Combination With Steroids in Patients Undergoing Liver Transplantation and a Pharmacokinetics Study.
Brief Title: A Study to Compare the Efficacy and Safety of FK506MR vs Prograf® in Patients Undergoing Liver Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MR4LTxCN01
Record Dates: First submitted 2007-04-10; First posted 2007-04-12 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Liver Transplantation
Keywords: Liver Transplantation; Tacrolimus; Methylprednisolone; Prednisolone
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): In combination with steroids
  Interventions: Drug: Tacrolimus modified-release
- 2 (Active Comparator): In combination with steroids
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Tacrolimus modified-release — oral
  Other Names: Advagraf; FK506MR; MR4
  Arms: 1
Drug: Prograf — oral
  Other Names: tacrolimus; FK506
  Arms: 2

SUMMARY:
The patients about to undergo liver transplantation will be randomized to one of the following two group:

Group FK506MR: FK506MR/steroid; Group Prograf® : Prograf® /steroid The treatment period is 3 months(12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent with the date of the patient must be obtained.
* Patient between 18-70 years of age receiving the primary liver.
* Female patients must have a negative pregnancy test prior to the enrolment.
* Female patients of child bearing potential must agree to practice effective birth control during the study

Exclusion Criteria:

* Liver re-transplantation patients or received an organ transplantation other than a liver.
* Living-related liver transplantation patient.
* Patient has received an AB0 incompatible donor liver.
* Patient who needs antibody induction therapy.
* Patient with sever infection requiring treatment.
* Patient has any history of severe cardiovascular, respiratory disease; or history of malignancy, liver cancer not included.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Event rate of patients with acute rejections | 12 Weeks

SECONDARY OUTCOMES:
Incidence of and time to acute rejections | 12 Weeks
Overall frequency of acute rejections | 12 Weeks
Rate of patient and graft survival following transplantation. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Leng Xisheng, Principal Investigator — Department of Hepatobiliary surgery
Locations (5):
- China (5):
  - Beijing, Beijing Municipality
  - Guangzhou, Guangdong
  - Shanghai, Shanghai Municipality
  - Hangzhou, Zhejiang
  - Tianjin

IPD SHARING:
Plan to Share IPD: Undecided